CLINICAL TRIAL: NCT03590912
Title: Efficacy and Cost Analysis of Steroids in Treatment of Otitis Media With Effusion (OME) Compared to That of Combination of Antibiotic, Antihistaminic, and Nasal Decongestant
Brief Title: Efficacy and Cost Analysis of Steroids in Treatment of Otitis Media With Effusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lumbini Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 143
Record Dates: First submitted 2018-07-08; First posted 2018-07-18 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Otitis Media With Effusion
MeSH Terms: conditions — Otitis Media with Effusion | interventions — Mometasone Furoate; Anti-Bacterial Agents; Histamine Antagonists; levocetirizine; Nasal Decongestants; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Wait and watch (Group D) (No Intervention): Wait and watch for 1 month
- Mometasone spray (Group B) (Experimental): Standard dose of mometasone furoate nasal spray (one spray in each nostril once daily) for one month will be given
  Interventions: Drug: Mometasone 50 Mcg/Inh Nasal Spray
- antibiotic + histaminic + oxymetazoline drops (Group A) (Experimental): This group will receive oral cefpodoxime (10 mg/kg/day in two divided dose for a week) plus oral histaminics and oxymetazoline drops. Standard dose of oral histaminics (levocetirizine, 1.25 mg for age below six years, 2.5 mg for older age) for a month plus oxymetazoline nasal drops (Nasivion 0.025%) for two weeks will be given
  Interventions: Drug: Antibiotics + Antihistamine (levocetirizine) + Nasal decongestants (Oxymetazoline 0.025%)
- Oral steroid (Group C) (Experimental): Patients in this group will receive one mg/kg/day of oral prednisolone (Oral steroid) in two divided dose for a week followed by half mg/kg/day in two divided dose for next one week
  Interventions: Drug: Steroid Drug (prednisolone)

INTERVENTIONS:
Drug: Mometasone 50 Mcg/Inh Nasal Spray — One spray in each nostril once daily for one month
  Other Names: Metaspray nasal spray
  Arms: Mometasone spray (Group B)
Drug: Antibiotics + Antihistamine (levocetirizine) + Nasal decongestants (Oxymetazoline 0.025%) — Children in this group will be treated with antiboitics (syp cefpodoxime) at 10 mg/kg/day in two divided dose for a week, plus antihistamine and nasal decongestants. Oral levocetirizine (Syrup levocet 2.5 mg/5ml) 1.25 mg once daily for age up to six years, 2.5 mg once daily for elder children for a month, plus oxymetazoline (Nasivion) 0.025%, 4 drops twice daily for two weeks
  Other Names: Syp Cefpodoxime, Syrup levocetirizine 2.5mg/ml; Nasivion drop
  Arms: antibiotic + histaminic + oxymetazoline drops (Group A)
Drug: Steroid Drug (prednisolone) — This group will be treated with steroid drugs. Oral prednisolone, 1 mg/kg body weight daily in two divided dose for 1 week followed by half mg/kg/day in two divided dose for next one week.
  Arms: Oral steroid (Group C)

SUMMARY:
We intend to study the cost of treatment, efficacy and adverse effects for Otitis media with effusion.

DETAILED DESCRIPTION:
Treatment groups would be:

1. Cefpodoxime + oxymetaxoline drops + levocetirizine
2. Fluticasone intranasal spray
3. Short term oral steroids
4. Wait and watch

ELIGIBILITY:
Inclusion Criteria:

* history of mild ear ache or decreased hearing for three or more months, plus
* intact and immobile tympanic membrane by pneumatic otoscopy
* Type B tympanogram

Exclusion Criteria:

* any external ear condition that hampers visualization of tympanic membrane
* lost to follow up

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-02-16 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Non B type tympanogram | one month

SECONDARY OUTCOMES:
cost of treatment | one month
Adverse effects | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Lumbini Medical College, Tānsen, Palpa, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, Analytic Code
Time Frame: As soon as the article is published online. Life-long

REFERENCES:
- [Derived] Mulvaney CA, Galbraith K, Webster KE, Rana M, Connolly R, Tudor-Green B, Marom T, Daniel M, Venekamp RP, Schilder AG, MacKeith S. Topical and oral steroids for otitis media with effusion (OME) in children. Cochrane Database Syst Rev. 2023 Dec 13;12(12):CD015255. doi: 10.1002/14651858.CD015255.pub2. PMID 38088821